CLINICAL TRIAL: NCT07339124
Title: The Effect of Single Lung Ventilation Duration and Intraoperative Brain Oxygenation on Cognitive Function and Postoperative Pain in Geriatric Patients Undergoing Single Lung Ventilation; Prospective Observational Study
Brief Title: The Effect of Single Lung Ventilation Duration and Intraoperative Brain Oxygenation on Cognitive Function and Postoperative Pain in Geriatric Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Baldemir, Clinic Associate Professor, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 2024-BÇEK/426
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Anesthesia; Geriatric Anesthesia; One Lung Ventillation (OLV); POCD - Postoperative Cognitive Dysfunction; Postoperative Pain Management
Keywords: thoracic anesthesia; geriatric patients; cognitive function; one lung ventilation; cerebral oxygenation; postoperative pain
MeSH Terms: conditions — Postoperative Cognitive Complications; Pain, Postoperative | interventions — Cognitive Remediation; Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients over 65 years of age who will undergo single-lung ventilation with thoracotomy.: The duration of single-lung ventilation and cerebral oxygenation values administered to patients during the intraoperative period will be recorded. The effects of these values on postoperative cognitive function and pain will be analyzed using statistical methods.
  Interventions: Other: Cognitive Remediation; Other: Pain Medicine

INTERVENTIONS:
Other: Cognitive Remediation — One day before the operation, postoperative The Mini Mental Test (MMT) form will be completed by patients at 48 hours and on the 7th postoperative day
Other: Pain Medicine — Pain levels of patients at 1, 2, 4, 8, 16, and 24 hours after thoracotomy will be evaluated using the Visual Analog Scale (VAS)

SUMMARY:
One lung ventilation (OLV) is commonly used in thoracic surgery. Although the lack of ventilation of the lung in the surgical area (independent lung) during OLV redirects pulmonary blood flow to the dependent lung, shunt development is inevitable, and consequently, hypoxia is a frequently encountered condition. Therefore, one of the most important aspects that clinicians pay attention to during OLV is cerebral oxygen saturation in addition to peripheral oxygenation monitoring.

Studies have shown a correlation between decreased cerebral oxygen saturation and postoperative cognitive dysfunction (POCD). Patients undergoing OLV are also at risk of cerebral desaturation due to this non-physiological ventilation.

Patients undergoing OLV are at risk of cerebral oxygen desaturation. Therefore, in these patients, both cognitive dysfunction and changes in brain oxygenation can negatively affect pain-related centers, altering pain perception. Geriatric patients are particularly more affected by these negative effects. It is generally accepted by healthcare professionals specializing in pain management that the application of pain management should differ for elderly patients compared to younger patients. Analgesic dose adjustment should be done more carefully in geriatric patients. Increased sensitivity to opioids due to hypoxia can cause respiratory depression and increased analgesic effects. To avoid these, opioid dose adjustment is necessary in these patients. In conclusion, cerebral oxygen saturation measurement can be an effective method to detect cerebral oxygen desaturation, especially in the geriatric patient group. In this way, the effect of hypoxia caused by OLV on cerebral oxygen saturation can be detected early, and POCD can be limited. We believe that this situation can also contribute to effective postoperative pain management. This study aimed to investigate the effect of intraoperative brain oxygenation on cognitive function and postoperative pain in geriatric patients who underwent OLV.

MATERİAL AND METHODS This study will be conducted in accordance with the Helsinki Declaration and will take place at Health Sciences University Ankara Atatürk Sanatorium Training and Research Hospital . The study will be planned for geriatric patients over 65 years of age with a high school diploma or higher education level who have given informed consent and are scheduled for OLV with standard anesthesia monitoring. These patients, undergoing thoracic surgery via thoracotomy and who agree to participate in this study and sign an informed consent form, will be prospectively enrolled. A total of 30 patients will be included in our study. Preoperatively, patients will undergo standard monitoring including non-invasive arterial blood pressure, electrocardiography, and peripheral oxygen saturation (SpO2). Cerebral oxygenation of patients who have signed an informed consent form the day before will be recorded throughout the surgical procedure using probes placed on the forehead before the induction of anesthetic drugs.

The standard anesthesia and analgesia protocol that we routinely apply to patients will be applied throughout the surgery. Routine preoperative blood tests, age, height, weight, Body Mass Index (BMI), gender, diagnosis, preoperative comorbidities (hypertension, diabetes, coronary artery disease, chronic obstructive pulmonary disease, etc.), previous surgeries (any surgical procedure performed under general anesthesia before this study), American Society of Anesthesiologists ( ASA) score, and duration of surgery will be recorded for each patient. Hemodynamic data (systolic arterial pressure (SAP), diastolic arterial pressure (DAP), mean arterial pressure (MAP), pulse, SpO2, and cerebral oxygen saturation will be recorded before anesthesia induction, after induction, and at 5, 10, 20, 30, and 60 minutes after the start of OLV. These hemodynamic data will also be recorded at the end OLV and at the end of the operation. OLV duration, anesthesia duration, surgery duration, amount of fluid administered, urine output, and whether blood replacement was performed will be recorded. Visual Analog Scale (VAS) scores will be recorded at 1, 2, 4, 8, 16, and 24 hours postoperatively. Analgesic medications administered during the 24-hour postoperative period will also be recorded. VAS evaluation will be performed on a 100 mm scale, where 0: no pain and 100: maximum pain, indicating the patient's pain level. During this process, any possible side effects that may develop due to analgesic treatment will be recorded.

The Mini Mental Test (MMT) form will be completed by patients one day before surgery, 48 hours postoperatively, on the 7th day postoperatively. MMT consists of eleven items grouped under five main headings: Orientation, recording memory, attention and calculation, recall, and language, and is evaluated out of a total score of 30.

DETAILED DESCRIPTION:
H0: In geriatric patients with a high school diploma or higher education level who are undergoing single-lung ventilation, single-lung ventilation duration and intraoperative brain oxygenation have no effect on cognitive function.

H1: In geriatric patients with a high school diploma or higher education level who are undergoing single-lung ventilation, single-lung ventilation duration and intraoperative brain oxygenation have an effect on cognitive function.

H0: In geriatric patients with a high school diploma or higher education level who are undergoing single-lung ventilation, single-lung ventilation duration and intraoperative brain oxygenation have no effect on postoperative pain.

H1: In geriatric patients with a high school diploma or higher education level who are undergoing single-lung ventilation, single-lung ventilation duration and intraoperative brain oxygenation have an effect on postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 and over with a high school diploma or higher education
* Patients undergoing lung resection via thoracotomy (wedge resection, lingulectomy, segmentectomy, lobectomy, pneumonectomy)
* American Society of Anesthesiologists (ASA) score I-II-III,
* Body mass index (BMI) between 18-40 kg/m2,
* Patients undergoing surgery under general anesthesia will be included in the study.

Exclusion Criteria:

* Patients under 65 years of age, patients over 65 who are illiterate,
* Who have completed primary or secondary school,
* Patients with pre-existing cognitive impairment confirmed by preoperative Mini Mental State Examination (MMSE),
* Patients with a history of previously diagnosed mental illness, cerebrovascular disease, senile dementia, stroke,
* Patients using continuous anti-inflammatory/analgesic medications,
* Patients with preoperative chronic pain,
* Severe cardiovascular disease,
* Diagnosed neurological and psychiatric diseases,
* Patients allergic to the anesthetic and analgesic drugs to be administered,
* Patients with severe renal failure, gastrointestinal ulceration or severe asthma that prevents the administration of standard analgesia protocols,
* Patients undergoing surgery other than lung resection,
* Patients undergoing surgery with TIVA (total intravenous anesthesia) will be excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study will be conducted in accordance with the Helsinki Declaration and will take place at SBÜ Ankara Atatürk Sanatorium Training and Research Hospital after obtaining ethical committee approval. The study will be planned for geriatric patients over 65 years of age with a high school diploma or higher education level who have given informed consent and are scheduled for single-lung ventilation (TAV) with standard anesthesia monitoring
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Mini Mental Test Measurements | 24 hours before surgery, 48 hours after surgery, and on the 7th postoperative day, or 7 days before discharge, or immediately before discharge.
Mini Mental Test Measurements | 24 hours before surgery, 48 hours after surgery, and on the 7th postoperative day, or immediately before discharge if the discharge date is less than 7 days.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) scores | Visual Analog Scale (VAS) scores will be recorded at 1, 2, 4, 8, 16, and 24 hours postoperatively
  During VAS evaluation, the patient will be asked to indicate the location of their pain intensity on a 100 mm scale (0: no pain, 100: maximum pain),

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Öztürk Yalçın, Principal Investigator — ANKARA ATATURK SANATORİUM TRAİNİNG AND RESEARCH HOSPITAL
Locations (1):
- Ankara Ataturk Sanatorium Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No